CLINICAL TRIAL: NCT04769479
Title: A Single Dose Study to Evaluate the Pharmacokinetics of Acoramidis Modified Release Tablet Formulations in Healthy Subjects
Brief Title: A Single Dose Study to Evaluate the Pharmacokinetics of Acoramidis Modified Release Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG10-006
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-03

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — attruby

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- acoramidis (Experimental)
  Interventions: Drug: acoramidis

INTERVENTIONS:
Drug: acoramidis — acoramidis
  Other Names: AG10

SUMMARY:
This is a single centre, open-label, 5-period study in healthy male and non-pregnant and non-lactating healthy female subjects.

DETAILED DESCRIPTION:
It is planned to enroll 14 subjects who will receive single oral doses of active IMP in a sequential manner over 5 periods, with a minimum of 7days between dosing in each period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females
* Body mass index (BMI) of 18.0 to 32.0kg/m² and a body weight>50kg as measured at screening
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must agree to adhere to the contraception requirements

Exclusion Criteria:

* Subjects who have received any IMP formulation in a clinical research study within the 90 days prior to Period 1, Day 1
* History of any drug or alcohol abuse in the past 2 years
* Subjects with pregnant or lactating partners
* Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are allowed.
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4g of paracetamol per day or HRT/hormonal contraception) in the 14 days before first IMP administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessments: Cmax | 72 hours
  Maximum Concentration (Cmax)
Pharmacokinetic Assessments: AUC | 72 hours
  Area under the plasma concentration-time curve (AUC)
Pharmacokinetic Assessments: Tmax | 72 hours
  Time to maximum concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MBChB, MRCS, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No